CLINICAL TRIAL: NCT00906776
Title: Randomised, Controlled, Clinical Study to Compare the Effect of a Combination of Enamel Matrix Proteins and Straumann Bone Ceramic With Autogenous Bone in Deep-wide Intrabony Defects
Brief Title: Emdogain and Straumann Bone Ceramic in Infrabony Defects
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty to recruit patients fulfilling inclusion criteria
Sponsor: Institut Straumann AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR 01/05
Record Dates: First submitted 2009-05-19; First posted 2009-05-21 (Estimated); Results first posted 2012-10-31 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-04

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Emdogain PLUS (Active Comparator): Straumann Emdogain in combination with Straumann BoneCeramic
  Interventions: Device: Emdogain PLUS
- Autogenous bone (Active Comparator): Autogenous bone from the patient
  Interventions: Device: Autogenous bone

INTERVENTIONS:
Device: Emdogain PLUS — Emdogain treatment followed by Straumann Bone Ceramic application during periodontal surgery
  Arms: Emdogain PLUS
Device: Autogenous bone — Autogenous bone application during periodontal surgery
  Arms: Autogenous bone

SUMMARY:
Randomised, controlled, clinical study to compare the effect of the combination of bone ceramic and enamel matrix proteins (test) versus autogenous bone graft alone (control) in the treatment of deep-wide intrabony defects

DETAILED DESCRIPTION:
30 subjects (15 test and 15 control) diagnosed with moderate to severe periodontitis (Armitage, 1999) will be enrolled in the study and randomized to either the test or the control group.

The surgical procedure shall be performed within 15 days from the baseline visit of the subjects and will be the same for both groups. In both groups, the flap is replaced subsequently.

In total 5 visits per patient are scheduled in this study. The total study duration for each patient should be 12 +/- 2 weeks.

The study devices Emdogain® and Straumann Bone Ceramic are CE-marked, and approved by the FDA.

One center in France will participate.

ELIGIBILITY:
Inclusion Criteria:

* Males and females must be at least 18 years and not more than 75 years of age
* The patient will have to be able to understand and sign the informed consent prior to starting the study.
* The patient also will have to have the ability and the willingness to comply with all study requirements.
* The patients will be in good general health without any systemic diseases.
* The teeth included in the study will be mandibular molars, maxillary and mandibular premolars, and canines.
* The patients will have to have at least one defect with pocket depth ≥ 5 mm.
* Intra-bony defects will have to have 1 or 2-wall morphology (at least 2/3 of the defect).
* Depth of the intrabony component of at least 3 mm
* The selected sites will have to have vertical intra-bony component ≥ 3 mm and an angle ≥ 30 degrees as assessed from standardized intra-oral radiographs.
* Oral hygiene parameters: Plaque Index (PI) ≤ 20 % and bleeding on probing (BoP) ≤ 20%

Exclusion Criteria:

* Heavy smokers: more than 20 cigarettes per day
* Mucosal diseases such as erosive lichen planus
* History of local radiation therapy
* Presence of oral lesions (such as ulceration, malignancy)
* Teeth with untreated endodontic or cardiologic problems
* Physical handicap that will interfere with patient's ability to exercise good oral hygiene on a regular basis.
* Patients presenting antibiotic treatment within the 3 months preceding the surgical procedure.
* Patients using anti-inflammatory drugs on a regular basis.
* Intra-bony defects with a 3-wall morphology.
* Intra-bony defects with furcation involvement.
* Incisors and maxillary molars, will be excluded.
* Alcoholism or chronically drug abuse causing systemic compromize
* Medical conditions requiring prolonged use of steroids
* Current pregnancy at the time of recruitment and/or breastfeeding women.
* Conditions or circumstances, in the opinion of the investigator, which could represent a general contra-indication for surgical procedure or would prevent completion of study participation or interfere with analysis of study results, such as history of non-compliance, or unreliability.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Bouchard, Prof, Principal Investigator — Rotschild Hospital
Locations (1):
- Hôtel-Dieu, Université Paris 7 Denis Diderot, Paris, France

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Emdogain PLUS | Autogenous Bone
Started | 11 | 8
Completed | 11 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Emdogain PLUS | Autogenous Bone | Total
Number analyzed (Participants) | 11 | 8 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.9 (8.9) | 31.9 (8.6) | 34.8 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinical Attachment Level (CAL)
Description: CAL is calculated as the sum of Probing Pocket Depth (PPD) and Recession (REC). PPD is measured using a periodontal probe from the gingival margin to the bottom of the pocket. REC is measured using a periodontal probe from the gingival margin to the cemento-enamel junction (CEJ).
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Emdogain PLUS | Autogenous Bone
Number analyzed (Participants) | 11 | 8
millimeters | -2.86 (1.43) | -2.44 (1.08)

2. Secondary Outcome: Change in Distance Between the Cementum-enamel-junction and the Base of the Vertical Bone Defect
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Emdogain PLUS | Autogenous Bone
Number analyzed (Participants) | 9 | 8
mm | -2.02 (1.80) | -2.13 (1.47)

3. Secondary Outcome: Change in Probing Pocket Depth (PPD)
Description: PPD is measured using a periodontal probe from the gingival margin to the bottom of the pocket.
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Emdogain PLUS | Autogenous Bone
Number analyzed (Participants) | 11 | 8
millimeters | -3.36 (1.42) | -2.75 (1.13)

4. Secondary Outcome: Change in Clinical Attachment Level (CAL)
Description: as for outcome 1
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Emdogain PLUS | Autogenous Bone
Number analyzed (Participants) | 11 | 8
mm | -2.44 (0.95) | -2.25 (1.10)

5. Secondary Outcome: Change in Probing Pocket Depth (PPD)
Description: PPD is measured using a periodontal probe from the gingival margin to the bottom of the pocket.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Emdogain PLUS | Autogenous Bone
Number analyzed (Participants) | 11 | 8
mm | -2.78 (1.18) | -2.56 (1.18)

6. Secondary Outcome: Change in Distance Between the Cementum-enamel-junction and the Base of the Vertical Bone Defect
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Emdogain PLUS | Autogenous Bone
Number analyzed (Participants) | 11 | 8
mm | -2.26 (1.99) | -2.29 (1.48)

ADVERSE EVENTS:
Arm/Group | Emdogain PLUS | Autogenous Bone
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/8
Other Adverse Events (participants affected / at risk) | 1/11 | 0/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Emdogain PLUS (N=11) | Autogenous Bone (N=8)
Pregnancy (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No